CLINICAL TRIAL: NCT03382886
Title: A Phase I Open Label Trial of a Combination of Nivolumab and Bevacizumab in Patients With Advanced and or Metastatic Hepatocellular Carcinoma
Brief Title: Nivolumab and Bevacizumab in Patients With Advanced and or Metastatic Hepatocellular Carcinoma
Acronym: NUANCE
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: PI decided to terminate due to low/slow accrual
Sponsor: University of Utah (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI103945
Record Dates: First submitted 2017-12-19; First posted 2017-12-26 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Hepatocellular Carcinoma
Keywords: Advanced and/or metastatic
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Nivolumab; Bevacizumab

STUDY DESIGN:
Intervention Model Description: This is an open label, phase I study to test for maximum tolerated dose (MTD) or recommended phase II dose (RP2D)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nivolumab and bevacizumab, all patients (Experimental)
  Interventions: Drug: Nivolumab; Drug: Bevacizumab

INTERVENTIONS:
Drug: Nivolumab — Nivolumab will be administered as a 240mg IV infusion given once every two weeks (+/- 3 days).
  Subjects will remain on study treatment for up to two years or until progression or excessive toxicity
  Other Names: OPDIVO
Drug: Bevacizumab — Bevacizumab will be administered as an IV infusion from 1-10mg/kg in accordance with the appropriate subject cohort being examined as described below:
  Dose level 1: 5 mg/kg intravenously once every two weeks Dose level 2: 10 mg/kg intravenously once every two weeks Dose level -1: 1 mg/kg intravenously once every two weeks
  Dosing is based on actual body weight. There is no dose adjustment for obese or frail individuals. Dosing is recalculated if patient weight changes by more than 10% as reviewed by the principal investigator.
  Subjects will remain on study treatment for up to two years or until progression or excessive toxicity

SUMMARY:
This is an open label, phase I study to test for maximum tolerated dose (MTD) or recommended phase II dose (RP2D) of the combination of nivolumab and bevacizumab. The study will use a 3+3 phase I study design using a fixed dose of nivolumab (240mg) and escalating doses of bevacizumab (1-10mg).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed unresectable or metastatic hepatocellular carcinoma. Confirmation either by histologic confirmation or accepted radiographic criteria.
* Received at least one line of therapy with a TKI (including, but not limited to sorafenib, lenvatinib, and/or regorafenib) with evidence of disease progression clinically or radiographically as deemed by investigator, or refused therapy with a TKI. No more than two lines of prior therapy are allowed.
* Measurable disease per RECIST1.1.
* Age ≥18 years.
* ECOG performance status of 0 to 1.
* Life expectancy ≥ 12 weeks.
* Childs Pugh A (5-6 points). Demonstrate adequate organ function as defined in the table below

Hematologic:

Absolute neutrophil count (ANC) ≥ 1.5 k/µL. Platelets ≥ 100 k/µL Hemoglobin ≥ 9 g/dL

Renal:

Creatinine < 2 × ULN OR

- Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines.

Exclusion Criteria:

* Prior treatment with anti-PD1 or anti-PD-L1 antibody therapy.
* Subjects with a prior history of DVT/PE, who have not been on stable doses of anticoagulation with low molecular weight heparin or oral anticoagulant for at least two weeks.
* History of arterial thromboembolic event in past 6 months (including CVA, MI).
* Systemic anti-cancer treatment within 2 weeks, all ongoing adverse events related to previous systemic anti-cancer therapy resolved to grade ≤1.
* Radiotherapy within 2 weeks of first dose of study medications.
* Major surgery within 6 weeks of first dose of study medications. Minor procedures (e.g. port placement, endoscopy with intervention) within 4 weeks of first dose of study medications.
* Presence of ≥ CTCAE grade 2 toxicity due to prior cancer therapy (except alopecia, peripheral neuropathy which are excluded if ≥ CTCAE grade 3).
* Medical condition that requires chronic systemic steroid therapy, or any other form of immunosuppressive medication.
* Active ongoing infection requiring therapy.
* Active HIV infection.
* History of severe hypersensitivity reaction to another monoclonal antibody.
* Active central nervous system metastases and/or carcinomatous meningitis (stable treated brain metastases not requiring steroids >4 weeks allowed).
* Cardiac conditions: class 3-4 New York Heart Association congestive heart failure, known baseline LVEF < 50%, transmural myocardial infarction, uncontrolled hypertension, angina pectoris requiring medication, clinically significant valvular disease, high-risk arrhythmia in the past 12 months.
* Any history of autoimmune disease requiring treatment in the past 5 years or felt to be at risk to reactivate autoimmune disease. Patients who are felt to no longer be at risk of activating a known autoimmune disease (e.g. type 1 diabetes, ulcerative colitis s/p complete colectomy, autoimmune thyroiditis s/p thyroidectomy or medical ablation, etc.) may be allowed to participate after discussion with the PI
* Pregnant, breast feeding, or planning to become pregnant.
* Women of childbearing potential (WOCBP) must agree to follow instructions for method(s) of contraception for the duration of study treatment with nivolumab and 5 months after the last dose of study treatment i.e., 30 days (duration of ovulatory cycle) plus the time required for the investigational drug to undergo approximately five half-lives. Contraception as described in section 7.3
* Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of study treatment with nivolumab and 7 months after the last dose of study treatment i.e., 90 days (duration of sperm turnover) plus the time required for the investigational drug to undergo approximately five half-lives. Contraception as described in section 7.3
* Received any live vaccine within the last 30 days.
* Other malignancy requiring treatment in the prior 2 years with the exception of locally treated squamous or basal cell carcinoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-04-11 (Actual); Primary Completion 2018-07-26 (Actual); Study Completion 2019-07-02 (Actual)

PRIMARY OUTCOMES:
Adverse Events that occur | Every 14 day cycle for up to 2 years - Patients are expected to be on treatment for an average of 6 months
  Investigate the safety and tolerability of 14-day cycles of nivolumab plus bevacizumab.
  Adverse events will be collected for each subject that received the study treatment combination.
Determine the maximum tolerated dose (MTD) or recommended phase 2 dose (RP2D) | The DLT period will begin at Cycle 1 Day 1 and continue through Cycle 1 Day 28 for each patient
  Determine the maximum tolerated dose (MTD) or recommended phase 2 dose (RP2D).
  Dose Limiting Toxicities (DLT) will define subsequent subject accrual and dose escalation

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | 3 years after treatment stops
  To examine the effect of the study treatment combination on the rate of progression-free survival (PFS).
  Subjects will have regular imaging scans to measure disease status and response will be defined by RECIST1.1.
Overall Survival | 3 years after treatment stops
  To examine the effect of the study treatment combination on the rate of overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Glynn W Gilcrease, MD, Principal Investigator — University of Utah
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States